CLINICAL TRIAL: NCT01352260
Title: Validation of Near-Infrared Spectroscopy for Neuromonitoring During Moderate Hypothermic Circulatory Arrest for Total Aortic Arch Replacement: A Comparison of Two Technologies With Jugular Venous Bulb Oximetry
Brief Title: Near-Infrared Spectroscopy Comparison Study
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: H-27855
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Total Aortic Arch Replacement
Keywords: Near Infrared Spectroscopy; Neuromonitoring; Aortic Arch Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Disease: Total Aortic Arch Replacement

SUMMARY:
The objective of this study is to validate Near-Infrared (NIRS) monitoring in patients undergoing circulatory arrest. This study will compare two-wavelength NIRS INVOS System, Somanetics; Troy, MI) with four-wavelength NIRS (Nonin Medical, Inc; Plymouth, MN) to determine which modality best correlates with jugular venous oxygen saturation

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent from patient or legally authorized representative before surgery
2. Adult patients 18-65 years of age
3. Presenting for elective or urgent total aortic arch repair under moderate hypothermic circulatory arrest (Nasopharyngeal temperature 20 - 24 ºC) with selective antegrade cerebral perfusion -

Exclusion Criteria:

1. Patients will be excluded from this study if they are age less than 18
2. Are undergoing an emergent procedure
3. Have a history of insulin-dependent diabetes mellitus
4. Have a history of stroke
5. Are undergoing a redo sternotomy during which major bleeding occurs necessitating transfusion of > 4 units of packed red blood cells prior to the institution of circulatory arrest
6. Patients in whom a left jugular venous bulb cannula cannot successfully be placed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Baylor College of Medicine and affiliated Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Linear correlation between absolute value of cerebral oxygen saturation (rSO2) compared to Jugular Venous Oxygen Saturation (SjvO2). Sensitivity and specificity to detect < 60% desaturation. | At the end of the surgical case approximately 6 to 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Wei Pan, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine and affiliated Hospitals, Houston, Texas, United States